CLINICAL TRIAL: NCT04598321
Title: BrUOG 390: Neoadjuvant Treatment With Talazoparib for Women With Newly Diagnosed, Advanced Ovarian Cancer Associated With a Mutation in BRCA1 or BRCA2 (mBRCA)
Brief Title: BrUOG 390: Neoadjuvant Treatment With Talazoparib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: termination of research grant agreement
Sponsor: Brown University (Other)
Collaborators: Pfizer (Industry); Lifespan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 390
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2022-12

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation; Ovarian Cancer; Fallopian Tube Cancer; High Grade Serous Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Planned Therapy (Experimental): Talazoparib monotherapy as 1 mg capsule orally on a daily basis for three cycles, defined as a 21-day period, prior to surgery. Volunteers will continue treatment to complete three cycles, unless disease progression or unacceptable toxicity occurs.Volunteers who complete neoadjuvant treatment with talazoparib should undergo surgical cytoreduction within three weeks of their last dose of talazoparib. All volunteers should then undergo standard of care adjuvant therapy using carboplatin and paclitaxel. For volunteers, who agree to continue talazoparib as maintenance therapy, treatment should begin three weeks (+/- 2 weeks) from the end of adjuvant chemotherapy or after cytoreductive surgery alone.
  Interventions: Drug: Talazoparib Oral Capsule

INTERVENTIONS:
Drug: Talazoparib Oral Capsule — An orally available PARP inhibitor for the treatment of advanced breast cancer with germline BRCA mutations.
  Other Names: Talzenna

SUMMARY:
Ovarian cancer is the most fatal gynecologic cancer; in the US alone an estimated 22,000 women will be diagnosed in 2019, with over 13,000 dying of the disease. Approximately half of epithelial ovarian cancers (EOC) exhibit defective DNA repair through alterations in the homologous recombination (HR) pathway, with 14% accounted for by germline mutations in BRCA genes (mBRCA); this goes up to about one in five (20%) women when one includes tumor-associated (somatic) mBRCA.The approach to women with mBRCA-associated ovarian cancer has heralded precision treatment in our field with the availability of PARP inhibitors. Now indicated as treatment for women with documented mBRCA (genomic or somatic), it also has shown significant benefits for women with recurrent EOC who respond to platinum-based therapy when administered as maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers must have clinical and radiographic evidence of newly detected FIGO stage II, III or IV epithelial ovarian, primary peritoneal or fallopian tube cancer, deemed by a gynecologic oncologist as not amenable to an R0 resection at presentation.
2. Institutional confirmation of Müllerian epithelial adenocarcinoma
3. Histologic epithelial cell types: high grade serous carcinoma, high grade endometrioid carcinoma, or a combination of these.
4. Documented mutation in BRCA1 or BRCA2 by genetic or commercial somatic testing. Reports will require submission at the time of enrollment.
5. Measurable disease as defined by RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or ≥ 20 mm when measured by chest x-ray. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI.14
6. Age ≥ 18
7. Adequate hematologic function determined within 28 days of consent as follows:

   * ANC greater than or equal to 1,500/mcl. NOTE: ANC cannot have been induced by granulocyte colony stimulating factors.
   * Platelets greater than or equal to 100,000/mcl
   * Hemoglobin greater than 10 mg/dl (NOTE: While transfusions are permitted to achieve baseline hemoglobin level, patients must not have transfusion within 14 days prior to obtaining baseline screening labs)
8. Creatinine Clearance > 15 mL/min. (NOTE: Please see Section 6.2.1 for dosing requirements for patients with renal insufficiency)

   CrCl = (140- age in years) x weight in kg x 0.85/ 72 x serum creatinine in mg/ dL
9. Adequate hepatic function within 14 days prior to registration defined as follows:

   * Bilirubin ≤ 1.5 x ULN
   * ALT and AST < 2.5 x ULN
   * Alkaline phosphatase ≤ 2.5 x ULN
10. Neurologic function: Neuropathy (sensory and motor) less than or equal to CTCAE v5.0 Grade 1.
11. Ability to swallow and retain oral medication. Adequate gastrointestinal absorption with no use of parenteral nutrition within two weeks of trial enrollment and no evidence of bowel obstruction.
12. The volunteer must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

1. Suspected non-gynecologic malignancy, evidenced by tumor markers and/or histologic evaluation.
2. Prior history of other invasive malignancies, with the exception of nonmelanoma skin cancer and other specific malignancies as noted in Section 4.2.4 and Section 4.2.5 are excluded if there is any evidence of other malignancy being present within the last three years (2 years for breast cancer, see Section 4.2.4). Volunteers are also excluded if their previous cancer treatment contraindicates this protocol therapy.
3. Prior chemotherapy for any abdominal or pelvic tumor within the last three years is excluded. Volunteers may have received prior adjuvant chemotherapy and radiotherapy for localized breast cancer, provided that it was completed more than 2 years prior to registration, the volunteer remains free of recurrent or metastatic disease and hormonal therapy has been discontinued.
4. Prior radiotherapy to any portion of the abdominal cavity or pelvis or thoracic cavity within the last three years are excluded. Prior radiation for localized cancer of the head and neck or skin is permitted, provided that it was completed more than three years prior to registration, and the volunteer remains free of recurrent or metastatic disease.
5. Synchronous primary endometrial cancer, or a past history of primary endometrial cancer, unless all of the following conditions are met: Stage not greater than I-A, grade 1 or 2, no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including serous, clear cell or other FIGO grade 3 lesions.
6. Severe, active co-morbidity defined as follows:

   * Chronic or current active infectious disease requiring systemic antibiotics, antifungal or antiviral treatment
   * Known brain or central nervous system metastases or history of uncontrolled seizures
   * Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months from enrollment, New York Heart Association Class III or IV congestive heart failure, and serious arrhythmia requiring medication (this does not include asymptomatic atrial fibrillation with controlled ventricular rate).
   * Partial or complete gastrointestinal obstruction
7. Volunteers who are not candidates for major abdominal surgery due to known medical comorbidities.
8. Volunteers with any condition that in the judgment of the investigator would jeopardize safety or volunteer compliance with the protocol.
9. Concurrent anticancer therapy (e.g. chemotherapy, radiation therapy, biologic therapy, immunotherapy, hormonal therapy, investigational therapy).
10. Receipt of an investigational study drug for any indication within 30 days or 5 half-lives (whichever is longer) prior to Day 1 of protocol therapy.
11. Prior exposure to a PARP inhibitor.
12. People of child-bearing potential (WOCB). This includes:

    * Any volunteer who has experienced menarche and who has not undergone surgical sterilization (hysterectomy and/or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12-month amenorrhea in a woman over 45 in the absence of other biological or physiological causes.
    * Volunteers who are pregnant or nursing. Volunteers must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 7 months after completing therapy.

    People with an intact uterus and ovaries must have a screening negative serum or urine pregnancy test within 14 days of registration. A second pregnancy test must be done within 24 hours prior to the start of the first cycle of study treatment
13. Potent P-gp inhibitors that result in ≥ 2-fold increase in the exposure of an in vivo probe P-gp substrate, including: amiodarone, carvedilol, clarithromycin, cobicistat, dronedarone, erythromycin, glecaprevir/pibrentasvir, indinavir, itraconazole, ketoconazole, lapatinib, lopinavir, propafenone, quinidine, ranolazine, ritonavir, saquinavir, sofosbuvir/velpatasvir/voxilaprevir, telaprevir, tipranavir, valspodar and verapamil.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female sex at birth.
Enrollment: 1 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don S Dizon, MD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - Women & Infants Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Planned Therapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Planned Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 62 [62 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Determine the Preliminary Effectiveness of Talazorparib
Description: Define the proportion of volunteers completing the planned 9 weeks of treatment without disease progression.
Time Frame: First 9 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Planned Therapy
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Feasibility of the Trial Design.
Description: Define whether 30 volunteers can successfully be enrolled within 2 years within participating institutions.
Time Frame: First 2 years of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Planned Therapy
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: From the time a signed and dated ICF was obtained until 30 days after the last treatment, approximately 8 months.
Arm/Group | Planned Therapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Planned Therapy (N=1)
Small intestinal obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Planned Therapy (N=1)
Anemia (Blood and lymphatic system disorders) | 1
Endocrine disorders, other (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Ileal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT04598321/Prot_SAP_ICF_000.pdf